CLINICAL TRIAL: NCT06787209
Title: Effects of a Hip Flexor and Extensor Muscle Training Program in Individuals with Chronic Mechanical Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lucía Pilar Vicente Pina (Other)
Responsible Party: Sponsor-Investigator, Lucía Pilar Vicente Pina, Trainee Researcher at the Department of Physiatry and Nursing, Universidad de Zaragoza
Organization: Universidad de Zaragoza (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI24/303
Record Dates: First submitted 2024-10-21; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: Chronic low back pain; hip flexors; Exercise therapy; lumbopelvic function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Public healthcare treatment (Active Comparator): Participants will receive four weeks of convetional active treatment for chronic low back pain at the healthcare center.
  Interventions: Behavioral: generic health care
- Program to improve lumbopelvic function (Experimental): The program will consist of a mixed model of in-person and home-based sessions. In-person sessions will be once a week and supervised by a physiotherapist. After each session participants will be encourage to replicate that session at home as many times as possible. Each session will include a warm-up, a strengthening phase, and a stretching phase. The strengthening part will be performed using a low-load methodology, which is the best alternative for home-based training. Specifically, the training will focus on stretching the hip flexors and strengthening the hip extensors.
  Interventions: Behavioral: Program to improve lumbopelvic function.

INTERVENTIONS:
Behavioral: Program to improve lumbopelvic function. — Each individual will receive a weekly session log at the start of the intervention, allowing them to record the total number of sessions performed between in-person visits and the perceived exertion.
  In the strengthening phase, both compound and isolated exercises will be performed. These exercises will be of low intensity and maintained for prolonged periods until the patient reaches fatigue or can no longer perform the repetitions correctly. If the patient reaches 40 repetitions, the exercise will be progressed in difficulty. The patient will have one minute of rest after each set.
  Each session will include a total of 4 sets focused on the gluteal muscles The speed of execution for each repetition will be between 4-6 seconds. After the strengthening phase, three unilateral static stretches targeting the hip flexors will be performed, each lasting one minute.
  The entire program will be performed using bodyweight exercises and adapted exercises that can be done at home.
  Arms: Program to improve lumbopelvic function
Behavioral: generic health care — The patients will receive 10 physiotherapy sessions at the health center throughout 4 weeks.They will be taught active exercises and undergo passive therapies to address their low back pain. Each session will last approximately 30 minutes.
  The intervention will therefore be variable depending on the assigned physiotherapist, as there is no standardized protocol for action.
  Arms: Public healthcare treatment

SUMMARY:
The goal of this clinical trial is to evaluate the effect of a physiotherapy intervention program in the lumbopelvic area in chronic low back pain patients. The main questions it aims to answer are:

1. Is a specific stretching and strengthening program for the hip musculature beneficial for function and symptom reduction in patients with non-specific chronic low back ain?
2. Are patients who have greater hip extension dysfunction going to benefit more from a specific program of stretching and strengthening of hip muscles?
3. Are there more alteration in pelvis alignement and movement in standig position compared to seated position in those patiens with lesser hip range of movement?
4. Are patiens with lesser hip range of movement going to show more dysfunction in the lumbopelvic region?

Participants will:

* Visit the physiotherapy clinic once a week to complete the therapeutic exercise session.
* Repeat the session in their houses if its possible between 3 or 4 times a week and record the number of days they repeat the session at home.
* Answer some questionaires at the begining of the intervention, after 4 weeks, a month and three months.

DETAILED DESCRIPTION:
This study aims to enhance healthcare interventions for chronic low back pain, focusing specifically on patients whose pain may be linked to restricted hip extension mobility. Patients will be referred from the healthcare system to the physiotherapy center, where the principal investigator, Lucía Vicente, will randomize participants into either the intervention or control group. Each participant will complete an initial evaluation at the start of the intervention and again after 4 weeks. Additional questionnaires will be administered one and three months post-intervention. Pelvic movement changes will also be tracked before each in-person session. The program will focus on strengthening the pelvic muscles, particularly by targeting hip extensor strengthening and hip flexor stretching.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 and less than 70 years.
* Low back pain lasting more than 3 months defined as: "Pain or discomfort localized below the costal margin and above the gluteal fold, with or without referred pain to the leg."
* Low back pain with a mechanical component.
* Signed informed consent prior to participation in the study.

Exclusion Criteria:

* A specific cause for their low back pain (trauma, spondylolisthesis, vertebral fractures, etc.), have undergone any surgical procedures on the spine or hip, or have other diseases or conditions (neurological issues, joint replacements, etc.).
* Cognitive impairment and inability to comprehend.
* Injections in the last 6 months or physiotherapy treatment in the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Hip flexors range of movement | From the enrollement to the end of the treatment at 4 weeks
  Range of motion of the hip flexors will be assessed using the Modified Thomas Test, also recording the body area where the sensation of stretch is felt, as well as the intensity.
Hip flexors range of movement | From the enrollement to the end of the treatment at 4 weeks
  Range of motion of the hip flexors will be assessed using The modified Ober test, also recording the body area where the sensation of tension or stretch is felt, as well as the intensity.

SECONDARY OUTCOMES:
Pain | From enrollment through the end of the 4-week treatment, and again one month after.
  Low back pain will be assessed using a visual analog scale (VAS). Information on average pain over the last 3 days, the maximum pain experienced, and the current pain level will be collected. The patient will mark their pain level with a line on scale ranging from 0 to 100 millimeters, where "0" represents no pain and "100" represents the worst imaginable pain, in relation to daytime pain (average VAS perceived over the last 3 days and at the present moment). Additionally, patients will be asked about the location and intensity of other symptoms using a Likert scale and a body map.
Oswestry Disability Index | From enrollment through the end of the 4-week treatment, and again one month after.
  It is a questionnaire composed of 10 categories: (1) pain intensity, (2) self-care, (3) lifting objects, (4) walking, (5) sitting, (6) standing, (7) sleeping, (8) sexual life, (9) social life, and (10) traveling. Each category consists of 6 items scored from 0 to 5, with a score of 0 on the first statement and 5 on the last. A mark at the highest levels indicates that the person is in worse condition. The questionnaire includes an additional question about previous treatments. If more than one response is selected, the highest score is considered. If all 10 sections are completed, the score is calculated as follows: the maximum score for the 10 sections is 50 points. If all sections are completed, this number is converted into a percentage with a total of 100. The Spanish version of the questionnaire shows good reliability and validity with an ICC between 0.89-0.97 and was validated in Spanish.
Pelvis saggital movement | From the enrollement to the end of the treatment at 4 weeks. For participants enrolled in the program to improve lumbopelvic function, this assessment will also be performed after each physiotherapy session.
  The pelvic movement will be recorded in video format in the sagittal plane for each patient in both standing and sitting positions with 45° of hip flexion. In each measurement it will be registered the range of movemento of the pelvis. The movement consist of the total range of anterior and posterior rotation of the pelvis.
Pain during pelvic tilting | From the enrollement to the end of the treatment at 4 weeks. For participants enrolled in the program to improve lumbopelvic function, this assessment will also be performed after each physiotherapy session.
  Pain during pelvic tilting will be assessed using a visual analog scale (VAS). The patient will mark their pain level with a line on scale ranging from 0 to 100 millimeters, where "0" represents no pain and "100" represents the worst imaginable pain. Additionally, patients will be asked about the location using a a body map and also the movement phase where the pain appears or is at its worst.

OTHER OUTCOMES:
Force in Newtons by a Maximum voluntary isometric contraction (MVIC) test | From the enrollement to the end of the treatment at 4 weeks
  A maximum voluntary isometric contraction (MVIC) test will be performed for the biceps femoris, gluteus maximus and tensor fasciae latae using a load cell.
Dynamic Activation Assessment during walking | From the enrollement to the end of the treatment at 4 weeks
  To assess dynamic activation, a gait test will be used. The gait test will involve walking on a treadmill for one minute at a comfortable speed, chosen by each patient. Two repetitions will be performed. Additionally, each subject will have an adaptation period to ensure they feel comfortable during the test.
  To assess activation, internal oblique, lumbar multifidus, gluteus maximus, and tensor fasciae lataewill be recorded simultaneously.
  The total percentage of activation for each muscle during the central 30 seconds of the test will be calculated.
  In addition, the speed achieved by each participant will also be recorded.
Anthropometric Data (weight) | From the enrollement to the end of the treatment at 4 weeks
  Weight in kq using the Tanita TBF-300, Amsterdam, Belgium
Sleep Quality | From the enrollement to the end of the treatment at 4 weeks, and a month after.
  The MOS Sleep Scale (Sleep Scale from the Medical Outcomes Study) will be used, which has proven to be a valid and reliable tool.
Kinesiophobia | From enrollment through the end of the 4-week treatment, and again one month after.
  The Tampa Scale for Kinesiophobia-11 (TSK-11) is a self-administered questionnaire recommended by the clinical guidelines for neuropathic pain assessment to measure fear of movement. It consists of 11 items assessing two factors: Activity Avoidance and Fear of Harm. Each item is rated on a 4-point Likert scale ranging from strongly disagree to strongly agree. High scores indicate a greater degree of kinesiophobia.
Sensitization Questionnaire | From enrollment through the end of the 4-week treatment, and again one month after.
  This instrument measures symptoms related to central sensitization syndromes. Part A assesses 25 common symptoms related to central sensitization syndromes, with a total score ranging from 0 to 100. Part B (not scored) asks if the participant has been diagnosed with one or more specific conditions, including seven different central sensitization syndromes.
Pain Catastrophizing Scale (PCS) | From the enrollement to the end of the treatment at 4 weeks, and a month after.
  The PCS is a 13-item self-administered scale and one of the most widely used to assess pain catastrophizing. It comprises three dimensions: a) rumination, b) magnification, and c) helplessness. The theoretical range of the scale is between 13 and 62, with lower scores indicating low catastrophizing and higher scores indicating severe catastrophizing.
COOP-WONCA Charts | From the enrollement to the end of the treatment at 4 weeks
  These charts assess health-related quality of life or perceived health. The questionnaire consists of 6 charts on health status and a total of 7 questions with five possible answers.
Mental Health Status | From enrollment through the end of the 4-week treatment, and again one month after.
  Assessed using the validated Spanish version of the GHQ-12 (General Health Questionnaire), which evaluates overall psychological well-being to detect non-psychotic psychiatric problems.The total score ranges from 0 to 12, with higher scores indicating poorer mental health. A cutoff score above 3 suggests psychological distress.
Emotional and Social Support | From enrollment through the end of the 4-week treatment, and again one month after.
  Assessed using the DUKE-UNC-11 (Duke-UNC Functional Social Support Questionnaire).The total score ranges from 11 to 55, categorizing the individual's perceived social support as "low" (below 32) or "normal" (32 or above)
Dynamic Activation Assessment durign Pelvic tilt | From the enrollement to the end of the treatment at 4 weeks
  To assess dynamic activation, a pelvic mobility test will be used. To assess activation, internal oblique, lumbar multifidus, gluteus maximus, and tensor fasciae lataewill be recorded simultaneously.
  The pelvic mobility test will be the same one used to analyze biomechanical variables. It will consist of an assessment in both standing and seated positions at 45° flexion, during which the electromyographic activity of the aforementioned muscles will be recorded simultaneously. The percentage of muscle activation during anterior and posterior pelvic tilts will be calculated in both standing and seated positions.
Walking speed | From the enrollement to the end of the treatment at 4 weeks
  The gait test will involve walking on a treadmill for one minute at a comfortable speed chosen by each patient. Two repetitions will be performed. Additionally, each subject will have an adaptation period to ensure they feel comfortable during the test.
  The speed achieved by each participant will be recorded, as lower speeds are associated with protective mechanisms.
Muscle activity during a Maximum voluntary isometric contraction (MVIC) test | From the enrollement to the end of the treatment at 4 weeks
  A maximum voluntary isometric contraction (MVIC) test will be performed for the biceps femoris, gluteus maximus, lumbar multifidus, internal oblique , and tensor fasciae latae using a wireless surface electromyography (EMG) system (Trigno Avanti, Delsys, Natick, USA).
  The electrode placement will follow the SENIAM recommendations. Each test will be performed for 3 seconds with 20 secons rest. The percentage of activation and peak activation will be recorded for each test.
Anthropometric Data (Height) | At the begining of the enrollement
  Height in centimeters using a stadiometer.
Body composition, percentage of Fat mass | From the enrollement to the end of the treatment at 4 weeks
  Fat mass wil be assessed using the Tanita bioelectrical impedance analyzer, with results expressed as a percentage relative to total body mass.
waist circumference | From the enrollement to the end of the treatment at 4 weeks
  waist circumference using a non-extensible plastic tape (TECSYMP Instruments: 0-2 m).
Body composition, percentage of muscle mass | From the enrollement to the end of the treatment at 4 weeks
  Muscle mass wil be assessed using the Tanita bioelectrical impedance analyzer, with results expressed as a percentage relative to total body mass.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Clinico de Fisioterapia OMT, Zaragoza, Zaragoza, Spain

REFERENCES:
- [Background] Iversen VM, Norum M, Schoenfeld BJ, Fimland MS. No Time to Lift? Designing Time-Efficient Training Programs for Strength and Hypertrophy: A Narrative Review. Sports Med. 2021 Oct;51(10):2079-2095. doi: 10.1007/s40279-021-01490-1. Epub 2021 Jun 14. PMID 34125411
- [Background] Jimenez-Del-Barrio S, Mingo-Gomez MT, Estebanez-de-Miguel E, Saiz-Cantero E, Del-Salvador-Miguelez AI, Ceballos-Laita L. Adaptations in pelvis, hip and knee kinematics during gait and muscle extensibility in low back pain patients: A cross-sectional study. J Back Musculoskelet Rehabil. 2020;33(1):49-56. doi: 10.3233/BMR-191528. PMID 31403939
- [Background] Zafereo J, Devanna R, Mulligan E, Wang-Price S. Hip stiffness patterns in lumbar flexion- or extension-based movement syndromes. Arch Phys Med Rehabil. 2015 Feb;96(2):292-7. doi: 10.1016/j.apmr.2014.09.023. Epub 2014 Oct 13. PMID 25312581
- [Background] Vigotsky AD, Lehman GJ, Contreras B, Beardsley C, Chung B, Feser EH. Acute effects of anterior thigh foam rolling on hip angle, knee angle, and rectus femoris length in the modified Thomas test. PeerJ. 2015 Sep 24;3:e1281. doi: 10.7717/peerj.1281. eCollection 2015. PMID 26421244